CLINICAL TRIAL: NCT03370679
Title: The Prognostic Significance of Premature Ventricular Complexes in Patients Without Structural Heart Disease
Acronym: PULSE
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PULSE
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Premature Ventricular Complexes Multiple; Premature Ventricular Contraction
Keywords: Premature; Ventricular; Complexes; Beats; Prognosis
MeSH Terms: conditions — Ventricular Premature Complexes; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
With this project the investigators aim to investigate whether premature ventricular complexes (PVC) have a prognostic significance in persons without structural heart disease. Further the investigators look at the possible connection between PVC-morphology and clinical outcome and investigate whether advanced cardiac imaging-methods may identify subtle signs of heart disease in PVC-patients with normal findings at echocardiography.

DETAILED DESCRIPTION:
The PULSE project consists of four different studies:

* in study one the investigators include patients who are evaluated because of PVCs and have no signs of structural heart disease at echocardiography and exercise test. The investigators follow them (average follow-up time 3,5 years) to investigate if they have a higher mortality och cardiovascular morbidity than standard population
* in study two the investigators carry out a sub-group analysis of the population in study one to assess whether PVC:s different sites of origin (morphology) are related to the clinical outcome
* in study three the investigators include persons with a high PVC-burden (at least 10 000 PVC:s/day) and normal echocardiography. The included subjects undergo magnetic resonance (MR) to investigate whether it can identify signs of heart disease where standard echocardiography cannot

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with Premature Ventricular Complexes at Three major Hospitals in Stockholm, Sweden

Exclusion Criteria:

* History of Myocardial Infarction
* Undergone coronary arterty bypass grafting (CABG)
* Finding of Heart Failure at echocardiography
* Direct or indirect findings of coronary ischaemia at exercise test, coronary angiography or other equivalent examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Premature Ventricular Complexes treated at Three major hospitals in the Stockholm area (Danderyd Hospital, Karolinska Hospital and Södersjukhuset Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Average follow-up time 3,5 years
  Mortality compared with sex and age-matched control population. Data for Control population obtained via Socialstyrelsen (The Swedish Health Board)

SECONDARY OUTCOMES:
Cardiovascular morbidity | Average follow-up time 3,5 years
  Incidence of heart failure and myocardial infarction in the study population compared with age and sex-matched Controls. Control data obtained via Socialstyrelsen (The Swedish Health Board)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Scorza, MD, Principal Investigator — Karolinska Institutet - Danderyd Hospital
Locations (1):
- Hjärtkliniken Danderyds Sjukhus, Stockholm, Sweden